CLINICAL TRIAL: NCT00367133
Title: A Randomized Trial Comparing Intravitreal Triamcinolone Acetonide and Laser Photocoagulation for Diabetic Macular Edema
Brief Title: Intravitreal Triamcinolone Acetonide Versus Laser for Diabetic Macular Edema
Acronym: IVT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-105; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2006-08-03; First posted 2006-08-22 (Estimated); Results first posted 2010-07-09 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic; macular; edema; intravitreal; triamcinolone; laser; photocoagulation; DME
MeSH Terms: conditions — Edema | interventions — Lasers; Triamcinolone Acetonide; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Standard of care group: conventional treatment consisting of focal/grid photocoagulation.
  Interventions: Procedure: Standard of Care Group
- 2 (Experimental): Intravitreal injection of 1mg of triamcinolone acetonide
  Interventions: Drug: 1mg triamcinolone acetonide
- 3 (Experimental): Intravitreal injection of 4mg of triamcinolone acetonide
  Interventions: Drug: 4mg triamcinolone acetonide

INTERVENTIONS:
Procedure: Standard of Care Group — Standard of care group: conventional treatment consisting of focal/grid photocoagulation.
  Other Names: soc with laser; modified ETDRS photocoagulation
  Arms: 1
Drug: 1mg triamcinolone acetonide — Intravitreal injection of 1mg of triamcinolone acetonide at baseline. At each 4-month interval visit, the investigator will assess whether persistent or recurrent DME is present that warrants retreatment with the randomization assigned treatment. Retreatment, when indicated, will be performed within four weeks after the follow-up visit. Retreatment should not be performed sooner than 3.5 months from the time of the last treatment.
  Other Names: corticosteroid
  Arms: 2
Drug: 4mg triamcinolone acetonide — 4mg intravitreal triamcinolone acetonide injection at baseline. At each 4-month interval visit, the investigator will assess whether persistent or recurrent DME is present that warrants retreatment with the randomization assigned treatment. Retreatment, when indicated, will be performed within four weeks after the follow-up visit. Retreatment should not be performed sooner than 3.5 months from the time of the last treatment.
  Other Names: corticosteroid
  Arms: 3

SUMMARY:
The study involves the enrollment of patients over 18 years of age with diabetic macular edema(DME). Patients with one study eye will be randomly assigned (stratified by visual acuity and prior laser) with equal probability to one of the three treatment groups:

1. Laser photocoagulation
2. 1mg intravitreal triamcinolone acetonide injection
3. 4mg intravitreal triamcinolone acetonide injection

For patients with two study eyes (both eyes eligible at the time of randomization), the right eye (stratified by visual acuity and prior laser) will be randomly assigned with equal probabilities to one of the three treatment groups listed above. The left eye will be assigned to the alternative treatment (laser or triamcinolone). If the left eye is assigned to triamcinolone, then the dose (1mg or 4 mg) will be randomly assigned to the left eye with equal probability (stratified by visual acuity and prior laser).

The study drug, triamcinolone acetonide, has been manufactured as a sterile intravitreal injectable by Allergan. Study eyes assigned to an intravitreal triamcinolone injection will receive a dose of either 1mg or 4mg. There is no indication of which treatment regimen will be better.

Patients enrolled into the study will be followed for three years and will have study visits every 4 months after receiving their assigned study treatment. In addition, standard of care post-treatment visits will be performed at 4 weeks after each intravitreal injection.

DETAILED DESCRIPTION:
Diabetic retinopathy is a major cause of visual impairment in the United States. Diabetic macular edema (DME) is a manifestation of diabetic retinopathy that produces loss of central vision. Data from the Wisconsin Epidemiologic Study of Diabetic Retinopathy (WESDR) estimate that after 15 years of known diabetes, the prevalence of diabetic macular edema is approximately 20% in patients with type 1 diabetes mellitus (DM), 25% in patients with type 2 DM who are taking insulin, and 14% in patients with type 2 DM who do not take insulin.

In a review of three early studies concerning the natural history of diabetic macular edema, Ferris and Patz found that 53% of 135 eyes with diabetic macular edema, presumably all involving the center of the macula, lost two or more lines of visual acuity over a two year period. In the Early Treatment Diabetic Retinopathy Study (ETDRS), 33% of 221 untreated eyes available for follow-up at the 3-year visit, all with edema involving the center of the macula at baseline, had experienced a 15 or more letter decrease in visual acuity score (equivalent to a doubling of the visual angle, e.g., 20/25 to 20/50, and termed "moderate visual acuity loss").

In the ETDRS, focal/grid photocoagulation of eyes with clinically significant macular edema (CSME) reduced the risk of moderate visual loss by approximately 50% (from 24% to 12%, three years after initiation of treatment). Therefore, 12% of treated eyes developed moderate visual loss in spite of treatment. Furthermore, approximately 40% of treated eyes that had retinal thickening involving the center of the macula at baseline still had thickening involving the center at 12 months, as did 25% of treated eyes at 36 months.

Although several treatment modalities are currently under investigation, the only demonstrated means to reduce the risk of vision loss from diabetic macular edema are laser photocoagulation, as demonstrated by the ETDRS, and intensive glycemic control, as demonstrated by the Diabetes Control and Complications Trial (DCCT) and the United Kingdom Prospective Diabetes Study (UKPDS). In the DCCT, intensive glucose control reduced the risk of onset of diabetic macular edema by 23% compared with conventional treatment. Long-term follow-up of patients in the DCCT show a sustained effect of intensive glucose control, with a 58% risk reduction in the development of diabetic macular edema for the DCCT patients followed in the Epidemiology of Diabetes Interventions and Complications Study.

The frequency of an unsatisfactory outcome following laser photocoagulation in some eyes with diabetic macular edema has prompted interest in other treatment modalities. One such treatment is pars plana vitrectomy. These studies suggest that vitreomacular traction, or the vitreous itself, may play a role in increased retinal vascular permeability. Removal of the vitreous or relief of mechanical traction with vitrectomy and membrane stripping may be followed by substantial resolution of macular edema and corresponding improvement in visual acuity. However, this treatment may be applicable only to a specific subset of eyes with diabetic macular edema. It also requires a complex surgical intervention with its inherent risks, recovery time, and expense. Other treatment modalities such as pharmacologic therapy with oral protein kinase C inhibitors and antibodies targeted at vascular endothelial growth factor (VEGF) are under investigation. The use of intravitreal corticosteroids is another treatment modality that has generated recent interest.

The optimal dose of corticosteroid to maximize efficacy with minimum side effects is not known. A 4mg dose of Kenalog is principally being used in clinical practice. However, this dose has been used based on feasibility rather than scientific principles.

There is also experience using Kenalog doses of 1mg and 2mg. These doses anecdotally have been reported to reduce the macular edema. There is a rationale for using a dose lower than 4mg. Glucocorticoids bind to glucocorticoid receptors in the cell cytoplasm, and the steroid-receptor complex moves to the nucleus where it regulates gene expression. The steroid-receptor binding occurs with high affinity (low dissociation constant (Kd) which is on the order of 5 to 9 nanomolar). Complete saturation of all the receptors occurs about 20-fold higher levels, i.e., about 100-200 nanomolar. A 4mg dose of triamcinolone yields a final concentration of 7.5 millimolar, or nearly 10,000-fold more than the saturation dose. Thus, the effect of a 1mg dose may be equivalent to that of a 4mg dose, because compared to the 10,000-fold saturation, a 4-fold difference in dose is inconsequential. It is also possible that higher doses of corticosteroid could be less effective than lower doses due to down-regulation of the receptor. The steroid implant studies provide additional justification for evaluating a lower dose, a 0.5mg device which delivers only 0.5 micrograms per day has been observed to have a rapid effect in reducing macular edema.

There has been limited experience using doses greater than 4mg. Jonas' case series reported results using a 25mg dose. However, others have not been able to replicate this dose using the preparation procedure described by Jonas.

In the trial, 4mg and 1mg doses will be evaluated. The former will be used because it is the dose that is currently most commonly used in clinical practice and the latter because there is reasonable evidence for efficacy and the potential for lower risk. Although there is good reason to believe that a 1mg dose will reduce the macular edema, it is possible that the retreatment rate will be higher with this dose compared with 4mg since the latter will remain active in the eye for a longer duration than the former. Insufficient data are available to warrant evaluating a dose higher than 4mg at this time.

ELIGIBILITY:
To be eligible, the following inclusion criteria must be met:

1. Age ≥18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2)
3. Able and willing to provide informed consent.
4. Patient understands that (1) if both eyes are eligible at the time of randomization, one eye will receive intravitreal triamcinolone acetonide and one eye will receive laser, and (2) if only one eye is eligible at the time of randomization and the fellow eye develops DME later, then the fellow eye will not receive intravitreal triamcinolone acetonide if the study eye received intravitreal triamcinolone acetonide (however, if the study eye was assigned to the laser group, then the fellow eye may be treated with the 4mg dose of the study intravitreal triamcinolone acetonide formulation, provided the eye assigned to laser has not received an intravitreal injection; such an eye will not be a "study eye" but since it is receiving study drug, it will be followed for adverse effects).

Exclusion Criteria

A patient is not eligible if any of the following exclusion criteria are present:

7. History of chronic renal failure requiring dialysis or kidney transplant.

8. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control). Note: Patients in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.

9. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at the time of study entry.

10. Known allergy to any corticosteroid or any component of the delivery vehicle.

11. History of systemic (e.g., oral, IV, IM, epidural, bursal) corticosteroids within 4 months prior to randomization or topical, rectal, or inhaled corticosteroids in current use more than 2 times per week.

12. Patient is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 3 years of the study.

13. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). Note: If blood pressure is brought below 180/110 by anti-hypertensive treatment, patient can become eligible.

Study Eye Eligibility

Inclusion

1. Best corrected Electronic-Early Treatment Diabetic Retinopathy Study (e-ETDRS) visual acuity score of ≥ 24 letters (i.e., 20/320 or better) and ≤73 letters (i.e., 20/40 or worse).
2. Definite retinal thickening due to diabetic macular edema based on clinical exam involving the center of the macula.
3. Mean retinal thickness on two Optical Coherence Tomography (OCT) measurements ≥250 microns in the central subfield.
4. Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photographs.

   Exclusion
5. Macular edema is considered to be due to a cause other than diabetic macular edema.
6. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, nonretinal condition).
7. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.)
8. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
9. History of prior treatment with intravitreal corticosteroids.
10. History of peribulbar steroid injection within 6 months prior to randomization.
11. History of focal/grid macular photocoagulation within 15 weeks (3.5 months) prior to randomization.Note: Patients are not required to have had prior macular photocoagulation to be enrolled. If prior macular photocoagulation has been performed, the investigator should believe that the patient may possibly benefit from additional photocoagulation.
12. History of panretinal scatter photocoagulation (PRP) within 4 months prior to randomization.
13. Anticipated need for PRP in the 4 months following randomization.
14. History of prior pars plana vitrectomy.
15. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 6 months following randomization.
16. History of YAG capsulotomy performed within 2 months prior to randomization.
17. Intraocular pressure ≥25 mmHg.
18. History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma.) Note: Angle-closure glaucoma is not an exclusion. A history of ocular hypertension is not an exclusion as long as (1) intraocular pressure (IOP) is <25 mm Hg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's diabetic retinopathy), and (4) the optic disc does not appear glaucomatous. If the intraocular pressure is 22 to <25 mm Hg, then the above criteria for ocular hypertension eligibility must be met.
19. History of steroid-induced intraocular pressure elevation that required IOP-lowering treatment.
20. History of prior herpetic ocular infection.
21. Exam evidence of ocular toxoplasmosis.
22. Aphakia.
23. Exam evidence of pseudoexfoliation.
24. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

In patients with only one eye meeting criteria to be a study eye at the time of randomization, the fellow eye must meet the following criteria:

1. Best corrected e-ETDRS visual acuity score ≥19 letters (i.e., 20/400 or better).
2. No prior treatment with intravitreal corticosteroids.
3. Intraocular pressure < 25 mmHg.
4. No history of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma.)Note: Angle-closure glaucoma is not an exclusion. A history of ocular hypertension is not an exclusion as long as (1) intraocular pressure is <25 mmHg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's diabetic retinopathy), and (4) the optic disc does not appear glaucomatous. If the intraocular pressure is 22 to <25 mmHg, then the above criteria for ocular hypertension eligibility must be met.
5. No history of steroid-induced intraocular pressure elevation that required IOP-lowering treatment.
6. No exam evidence of pseudoexfoliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2004-07; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ip, M.D., Study Chair — University of Wisconsin Medical School
Locations (83):
- United States (83):
  - Jones Eye Institute/University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - SCPMG Regional Offices - Kaiser Permanente, Baldwin Park, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of California, Irvine, Irvine, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Doheny Eye Institute, Los Angeles, California
  - Jules Stein Eye Institute, Los Angeles, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - West Coast Retina Medical Group, Inc., San Francisco, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Denver Health Medical Center, Denver, Colorado
  - Eldorado Retina Associates, P.C., Louisville, Colorado
  - Connecticut Retina Consultants, New Haven, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - International Eye Center, Tampa, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Retina Associates of Hawaii, Inc., Honolulu, Hawaii
  - Retina Consultants of Hawaii, Inc., ‘Aiea, Hawaii
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Retina Associates, Joliet, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Vitreoretinal Consultants, Bangor, Maine
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Ophthalmological Institute at Johns Hopkins, Baltimore, Maryland
  - The Retina Group of Washington, Greenbelt, Maryland
  - Retina Consultants of Delmarva, P.A., Salisbury, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Associated Retinal Consultants, Grand Rapids, Michigan
  - Vision Research Foundation, Royal Oak, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis University Eye Institute, St Louis, Missouri
  - Barnes Retina Institute, St Louis, Missouri
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - University of Rochester, Rochester, New York
  - Retina Consultants, PLLC, Slingerlands, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - University of North Carolina, Dept. of Ophthalmology, Chapel Hill, North Carolina
  - Charlotte Eye Ear Nose and Throat Assoc, PA, Charlotte, North Carolina
  - Horizon Eye Care, PA, Charlotte, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - OSU Eye Physicians and Surgeons, LLC., Dublin, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Retina Consultants, Providence, Rhode Island
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - West Texas Retina Consultants P.A., Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - University of Texas Medical Branch, Dept of Ophthalmology and Visual Sciences, Galveston, Texas
  - Charles A. Garcia, PA & Associates, Houston, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Dept. of Ophthalmology, Madison, Wisconsin
  - Medical College of Wiconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Bhavsar AR, Ip MS, Glassman AR; DRCRnet and the SCORE Study Groups. The risk of endophthalmitis following intravitreal triamcinolone injection in the DRCRnet and SCORE clinical trials. Am J Ophthalmol. 2007 Sep;144(3):454-6. doi: 10.1016/j.ajo.2007.04.011. PMID 17765429
- [Result] Ip MS, Bressler SB, Antoszyk AN, Flaxel CJ, Kim JE, Friedman SM, Qin H; Diabetic Retinopathy Clinical Research Network. A randomized trial comparing intravitreal triamcinolone and focal/grid photocoagulation for diabetic macular edema: baseline features. Retina. 2008 Jul-Aug;28(7):919-30. doi: 10.1097/IAE.0b013e31818144a7. PMID 18698292
- [Result] Diabetic Retinopathy Clinical Research Network. A randomized trial comparing intravitreal triamcinolone acetonide and focal/grid photocoagulation for diabetic macular edema. Ophthalmology. 2008 Sep;115(9):1447-9, 1449.e1-10. doi: 10.1016/j.ophtha.2008.06.015. Epub 2008 Jul 26. PMID 18662829
- [Result] Diabetic Retinopathy Clinical Research Network (DRCR.net); Beck RW, Edwards AR, Aiello LP, Bressler NM, Ferris F, Glassman AR, Hartnett E, Ip MS, Kim JE, Kollman C. Three-year follow-up of a randomized trial comparing focal/grid photocoagulation and intravitreal triamcinolone for diabetic macular edema. Arch Ophthalmol. 2009 Mar;127(3):245-51. doi: 10.1001/archophthalmol.2008.610. PMID 19273785
- [Result] Aiello LP, Edwards AR, Beck RW, Bressler NM, Davis MD, Ferris F, Glassman AR, Ip MS, Miller KM; Diabetic Retinopathy Clinical Research Network. Factors associated with improvement and worsening of visual acuity 2 years after focal/grid photocoagulation for diabetic macular edema. Ophthalmology. 2010 May;117(5):946-53. doi: 10.1016/j.ophtha.2009.10.002. Epub 2010 Feb 1. PMID 20122739
- [Result] Bressler NM, Edwards AR, Beck RW, Flaxel CJ, Glassman AR, Ip MS, Kollman C, Kuppermann BD, Stone TW; Diabetic Retinopathy Clinical Research Network. Exploratory analysis of diabetic retinopathy progression through 3 years in a randomized clinical trial that compares intravitreal triamcinolone acetonide with focal/grid photocoagulation. Arch Ophthalmol. 2009 Dec;127(12):1566-71. doi: 10.1001/archophthalmol.2009.308. PMID 20008708
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] Gangaputra S, Almukhtar T, Glassman AR, Aiello LP, Bressler N, Bressler SB, Danis RP, Davis MD; Diabetic Retinopathy Clinical Research Network. Comparison of film and digital fundus photographs in eyes of individuals with diabetes mellitus. Invest Ophthalmol Vis Sci. 2011 Aug 3;52(9):6168-73. doi: 10.1167/iovs.11-7321. PMID 21571677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-eight academic and community based sites across the United States recruited 693 subjects from May 2004 to July 2006.
Groups:
- Focal/Grid Laser Photocoagulation: Standard of care group: conventional treatment consisting of focal/grid photocoagulation.
- 1mg Intravitreal Triamcinolone: Intravitreal injection of 1mg of triamcinolone acetonide
- 4 mg Intravitreal Triamcinolone: Intravitreal injection of 4mg of triamcinolone acetonide
Period: 2 Years
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Started | 330 (Number of Eyes) | 256 (Number of Eyes) | 254 (Number of Eyes)
Completed | 272 | 220 | 205
Not Completed | 58 | 36 | 49
Not completed — Death | 20 | 12 | 12
Not completed — Dropped | 34 | 19 | 33
Not completed — Missed visit | 4 | 5 | 4
Period: 3 Years
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Started | 143 (Since trial ended early, includes only those with potential for 3 year follow-up -excludes deaths) | 116 (Since trial ended early, includes only those with potential for 3 year follow-up -excludes deaths) | 116 (Since trial ended early, includes only those with potential for 3 year follow-up -excludes deaths)
Completed | 115 | 93 | 98
Not Completed | 28 | 23 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone | Total
Number analyzed (Participants) | 330 | 256 | 254 | 840
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [57 to 69] | 63 [58 to 70] | 63 [57 to 69] | 63 [57 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 120 | 125 | 411
  Male | 164 | 136 | 129 | 429
Race/Ethnicity, Customized [Number; unit: participants]
  White | 243 | 186 | 183 | 612
  Black | 31 | 22 | 26 | 79
  Hispanic or Latino | 39 | 34 | 33 | 106
  Asian | 7 | 8 | 5 | 20
  American Indian/Alaskan Native | 2 | 2 | 2 | 6
  Native Hawaiian/other Pacific Islander | 1 | 0 | 1 | 2
  More than 1 race | 1 | 1 | 0 | 2
  Unknown/not reported | 6 | 3 | 4 | 13
Diabetes Type [Number; unit: Participants]
  Type 1 | 14 | 12 | 12 | 38
  Type 2 | 316 | 244 | 242 | 802
History of ocular hypertension [Number; unit: Eyes]
  Ocular Hypertension | 3 | 8 | 4 | 15
  No Ocular Hypertension | 327 | 248 | 250 | 825
Lens status phakic (clinical examination) [Number; unit: Eyes]
  Phakic | 262 | 203 | 197 | 662
  Pseudophakic | 68 | 53 | 57 | 178
OCT cystoid abnormality (questionable or definite) [Number; unit: Eyes]
  OCT cystoid abnormality (questionable or definite) | 315 | 243 | 246 | 804
  No Evidence | 12 | 9 | 6 | 27
  Missing/can not grade | 3 | 4 | 2 | 9
OCT subretinal fluid present (questionable or definite [Number; unit: Eyes]
  OCT subretinal fluid present | 94 | 64 | 61 | 219
  Missing (or ungradeable) | 1 | 4 | 1 | 6
  No OCT subretinal fluid present | 235 | 188 | 192 | 615
Prior Panretinal scatter photocoagulation [Number; unit: Eyes]
  Prior Panretinal scatter photocoagulation | 53 | 40 | 42 | 135
  No Prior Panretinal scatter photocoagulation | 277 | 216 | 212 | 705
Prior photocoagulation for diabetic macular edema [Number; unit: Eyes]
  Prior photocoagulation for DME | 198 | 154 | 158 | 510
  No Prior photocoagulation for DME | 132 | 102 | 96 | 330
Retinopathy severity (ETDRS severity scale) [Number; unit: Eyes] — Early Treatment Diabetic Retinopathy Study (ETDRS) scale. Retinopathy severity data missing for: 12, 8, 10 eyes in the Laser, 1mg and 4mg treatment groups, respectively.
  Eyes
    Microaneurysms only | 1 | 1 | 0 | 2
    Mild-moderately severe nonproliferative | 186 | 156 | 151 | 493
    Severe nonproliferative | 43 | 27 | 25 | 95
    Mild to moderate proliferative | 79 | 56 | 62 | 197
    High-risk proliferative | 9 | 8 | 6 | 23
    Missing (ungradeable) | 12 | 8 | 10 | 30
Visual Acuity Categorized by Randomization Strata [Number; unit: Eyes] — Letter score and approximate Snellen equivalent. Best score is 97, worst is 0.
  Eyes
    73-60 (20/32-2-20/62) | 189 | 149 | 149 | 487
    59-36 (<20/631-20/200) | 129 | 94 | 92 | 315
    35-24 (20/200-20/320) | 12 | 13 | 13 | 38
Central subfield thickness on OCT [Median (Inter-Quartile Range); unit: Microns] — Mean of two baseline scans. Mean CST <250 microns based on RC grading in 15, 7, and 5 eyes for laser, 1 mg, and 4 mg groups, respectively. Missing/ungradable optical coherence tomography or fundus photo data for 1, 2, and 1 eyes for laser, 1 mg, and 4 mg groups, respectively.
  Microns | 398 [329 to 505] | 405 [327 to 514] | 396 [323 to 484] | 400 [323 to 514]
Duration of Diabetes [Median (Inter-Quartile Range); unit: Years] | 15 [9 to 21] | 15 [9 to 21] | 16 [10 to 22] | 15 [9 to 22]
HbA1c [Median (Inter-Quartile Range); unit: Percentage] — Missing HbA1c data in 64, 46, and 50 in the laser, 1 mg, and 4 mg groups respectively
  Percentage | 7.5 [6.6 to 8.5] | 7.5 [6.8 to 8.4] | 7.6 [6.8 to 8.8] | 7.5 [6.6 to 8.8]
Intraocular pressure [Median (Inter-Quartile Range); unit: microns] | 16 [13 to 18] | 16 [13 to 18] | 16 [14 to 18] | 16 [13 to 18]
Retinal volume on OCT [Median (Inter-Quartile Range); unit: cubic millimetre] — Missing/ungradeable optical coherence tomography and fundus photo data for the laser, 1mg, and 4 mg groups respectively: 37, 36, 48.
  cubic millimetre | 9.2 [7.9 to 10.6] | 8.9 [7.8 to 10.5] | 8.9 [7.9 to 10.0] | 9.0 [7.8 to 10.6]
e-ETDRS visual acuity [Median (Inter-Quartile Range); unit: Letter Score] — Best corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. Best value on the scale 97, worst 0.
  Letter Score | 62 [53 to 67] | 62 [54 to 67] | 62 [52 to 67] | 62 [52 to 67]

OUTCOME MEASURES:

1. Primary Outcome: Change In Visual Acuity [Measured With Electronic-Early Treatment Diabetic Retinopathy Study (E-ETDRS)]Baseline to 2 Years.
Description: Change in best correct visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. A positive change denotes an improvement. Best value on the scale 97, worst 0.
Time Frame: Baseline to 2 Years
Population: The primary analysis included all randomized eyes and followed the intent-to-treat principle.
Measure: Mean (Standard Deviation); unit: Letter score
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 330 | 256 | 254
Letter score | 1 (17) | -2 (18) | -3 (22)
Statistical Analysis 1: Comparison: Focal/Grid Laser Photocoagulation vs 1mg Intravitreal Triamcinolone; P values for two group comparisons for difference in mean change; Test type: Superiority or Other; p = 0.02, ANCOVA; Repeated Measures Model. Adjusted for baseline visual acuity and prior photocoagulation; Accounted for correlated data from subjects with 2 study eyes
Statistical Analysis 2: Comparison: Focal/Grid Laser Photocoagulation vs 4 mg Intravitreal Triamcinolone; P Values for 2 group comparisons of difference in mean change; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 1mg Intravitreal Triamcinolone vs 4 mg Intravitreal Triamcinolone; P Values for 2 group comparisons of difference in mean change; Test type: Superiority or Other; p = 0.49, ANCOVA; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Central Subfield Thickness at 2 Years
Description: Median central subfield thickness at two-years. Optical coherence Tomography (OCT) images were obtained by a certified operator using the Zeiss Stratus OCT machine. If the automated thickness measurements were judged by the reading center to be inaccurate, center point thickness was measured manually, and this value was used to impute a value for the central subfield.
Time Frame: 2 Years
Population: Only subjects with an available Optical coherence tomography (OCT) at baseline and 2 years are included in the OCT analysis.
Measure: Median (Inter-Quartile Range); unit: Microns
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 261 | 207 | 193
Microns | 243 (148) [197 to 326] | 305 (167) [231 to 406] | 279 (160) [228 to 430]

3. Primary Outcome: Median Change in Visual Acuity Baseline to 2 Years
Description: Change in best correct visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. A positive change denotes an improvement.
Time Frame: Baseline to 2 Years
Population: The primary analysis included all randomized eyes and followed the intent-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: Letter score
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 330 | 256 | 254
Letter score | 4 [-6 to 11] | 1 [-11 to 9] | 2 [-11 to 11]

4. Primary Outcome: Distribution of Change in Visual Acuity Baseline to 2 Years
Description: Change in best correct visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method.
Time Frame: baseline to 2 years
Population: The primary analysis included all randomized eyes and followed the intent-to-treat principle
Measure: Number; unit: Percentage of Eyes
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 330 | 256 | 254
Percentage of Eyes
  >= 15 letter improvement | 18 | 14 | 17
  14 to 10 letter improvement | 13 | 11 | 11
  9 to 5 letter improvement | 16 | 14 | 15
  same +- 4 letters | 24 | 27 | 23
  5-9 letters worse | 10 | 9 | 6
  10-14 letters worse | 5 | 6 | 8
  >=15 letters worse | 14 | 20 | 20
Statistical Analysis 1: Comparison: Focal/Grid Laser Photocoagulation vs 1mg Intravitreal Triamcinolone; Proportion with 15-letter or more worsening; Test type: Superiority or Other; p = 0.03, GEE Repeated Measures; Hochberg procedure used to determine statistical significance
Statistical Analysis 2: Comparison: Focal/Grid Laser Photocoagulation vs 4 mg Intravitreal Triamcinolone; Proportion with 15-letter or more worsening; Test type: Superiority or Other; p = 0.01, GEE Repeated Measures; Hochberg procedure used to determine statistical significance
Statistical Analysis 3: Comparison: 1mg Intravitreal Triamcinolone vs 4 mg Intravitreal Triamcinolone; Proportion with 15-letter or more worsening; Test type: Superiority or Other; p = 0.82, GEE Repeated Measures; Hochberg procedure used to determine statistical significance

5. Secondary Outcome: Mean Change in Central Subfield Thickness Baseline to 2 Years
Description: Overall central subfield change from baseline. Optical coherence Tomography (OCT) images were obtained by a certified operator using the Zeiss Stratus OCT machine. The average of 2 baseline central subfield thickness measurements was used for analysis.If the automated thickness measurements were judged by the reading center to be inaccurate, center point thickness was measured manually, and this value was used to impute a value for the central subfield. Negative change denotes and improvement.
Time Frame: Baseline to 2 years
Population: Only subjects with available OCTs at baseline and 2 years are included in the OCT analysis.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 261 | 207 | 193
Microns | -139 (148) | -86 (167) | -77 (160)
Statistical Analysis 1: Comparison: Focal/Grid Laser Photocoagulation vs 1mg Intravitreal Triamcinolone; P value not adjusted for multiple comparisons; Test type: Superiority or Other; p < 0.001, ANCOVA; Repeated Measures Model. Accounted for correlated data from subjects with 2 study eyes; included baseline central subfield thickness as a covariate
Statistical Analysis 2: Comparison: Focal/Grid Laser Photocoagulation vs 4 mg Intravitreal Triamcinolone; P Value not adjusted for multiple comparisons; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 1mg Intravitreal Triamcinolone vs 4 mg Intravitreal Triamcinolone; P Values not adjusted for multiple comparisons; Test type: Superiority or Other; p = 0.91, ANCOVA; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Median Change in Central Subfield Thickness Baseline to 2 Years
Description: Overall central subfield change from baseline. Optical coherence Tomography (OCT) images were obtained by a certified operator using the Zeiss Stratus OCT machine. The average of 2 baseline central subfield thickness measurements was used for analysis.If the automated thickness measurements were judged by the reading center to be inaccurate, center point thickness was measured manually, and this value was used to impute a value for the central subfield. Negative change denotes an improvement.
Time Frame: Baseline to 2 Years
Population: Only subjects with an available OCT's at baseline and 2 years are included in the OCT analysis.
Measure: Median (Inter-Quartile Range); unit: Microns
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 261 | 207 | 193
Microns | -131 [-217 to -49] | -74 [-168 to -3] | -76 [-175 to 11]

7. Secondary Outcome: Overall Central Subfield Thickening Decreased by >=50% Baseline to 2 Years
Description: Overall central subfield change from baseline. Optical coherence Tomography (OCT) images were obtained by a certified operator using the Zeiss Stratus OCT machine. If the automated thickness measurements were judged by the reading center to be inaccurate, center point thickness was measured manually, and this value was used to impute a value for the central subfield.
Time Frame: Baseline to 2 Years
Population: Only subjects with available OCTs at baseline and 2 years are included in the OCT analysis.
Measure: Number; unit: Percentage of Eyes
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 261 | 207 | 193
Percentage of Eyes | 67 | 46 | 48
Statistical Analysis 1: Comparison: Focal/Grid Laser Photocoagulation vs 1mg Intravitreal Triamcinolone; P Values not adjusted for multiple comparisons; Test type: Superiority or Other; p < 0.001, GEE Repeated Measures; Accounted for correlated data from subjects with 2 study eyes; included baseline central subfield thickness as a covariate
Statistical Analysis 2: Comparison: Focal/Grid Laser Photocoagulation vs 4 mg Intravitreal Triamcinolone; P Values not adjusted for multiple comparisons; Test type: Superiority or Other; p < 0.001, GEE Repeated Measures; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: 1mg Intravitreal Triamcinolone vs 4 mg Intravitreal Triamcinolone; P Value not adjusted for multiple comparisons; Test type: Superiority or Other; p = 0.60, GEE Repeated Measures; [statistical method as in outcome 7, analysis 1]

8. Secondary Outcome: Central Subfield Thickness < 250 Microns at 2 Years
Description: as for outcome 7
Time Frame: 2 Years
Population: Only subjects with available OCTs at baseline and 2 years are included in the OCT analysis.
Measure: Number; unit: Percentage of Eyes
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 261 | 207 | 193
Percentage of Eyes | 53 | 34 | 38
Statistical Analysis 1: Comparison: Focal/Grid Laser Photocoagulation vs 1mg Intravitreal Triamcinolone; P Values not adjusted for multiple comparisons; Test type: Superiority or Other; p < 0.001, GEE Repeated Measures; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Focal/Grid Laser Photocoagulation vs 4 mg Intravitreal Triamcinolone; P Value not adjusted for statistical analysis; Test type: Superiority or Other; p < 0.001, GEE Repeated Measures; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: 1mg Intravitreal Triamcinolone vs 4 mg Intravitreal Triamcinolone; P Value not adjusted for statistical analysis; Test type: Superiority or Other; p = 0.55, GEE Repeated Measures; [statistical method as in outcome 7, analysis 1]

9. Secondary Outcome: Change in Visual Acuity From Baseline to 3 Years
Description: as for outcome 3
Time Frame: Baseline to 3 year
Population: The study discontinued early. Only subjects with 3 years data are included in 3 year analysis.
Measure: Mean (Standard Deviation); unit: Letter Score
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 115 | 93 | 98
Letter Score | 5 (17) | 0 (16) | 0 (21)

10. Secondary Outcome: Change in Visual Acuity From Baseline to 3 Years
Description: Change in best correct visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. A positive change denotes an improvement. Best Value on the scale=97, Worst Value=0
Time Frame: Baseline to 3 year
Population: The study discontinued early. Only subjects with 3 years data are included in 3 year analysis.
Measure: Median (Inter-Quartile Range); unit: Letter Score
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 115 | 93 | 98
Letter Score | 8 [-2 to 15] | 2 [-11 to 9] | 4 [-8 to 14]

11. Secondary Outcome: Distribution of Visual Acuity Change Baseline to 3 Years
Description: Change in best correct visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. A positive change denotes an improvement. Best value on the scale=97, worst=0
Time Frame: Baseline to 3 years
Population: The study discontinued early. Only subjects with 3 years data are included in 3 year analysis.
Measure: Number; unit: Percentage of Eyes
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 115 | 93 | 98
Percentage of Eyes
  >= 15 letters better | 26 | 20 | 21
  10-14 letters better | 18 | 4 | 16
  5-9 letters better | 18 | 17 | 9
  no change, + - 4 letters | 21 | 23 | 24
  5-9 letters worse | 4 | 10 | 6
  10-14 letters worse | 4 | 9 | 6
  >=15 letters worse | 8 | 17 | 16

12. Secondary Outcome: Central Subfield Thickness on Optical Coherence Tomography (OCT) at Three Years
Description: as for outcome 7
Time Frame: 3 years
Population: The study discontinued early. Only subjects with 3 years data are included in 3 year analysis.
Measure: Median (Inter-Quartile Range); unit: Microns
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 111 | 87 | 89
Microns | 211 [175 to 271] | 269 [210 to 299] | 248 [195 to 342]

13. Secondary Outcome: Change in Central Subfield Thickness on OCT Baseline to 3 Years
Description: as for outcome 6
Time Frame: Baseline to 3 years
Population: The study discontinued early. Only subjects with 3 years data are included in 3 year analysis.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 111 | 87 | 89
Microns | -175 (149) | -124 (184) | -126 (159)

14. Secondary Outcome: Change in Central Subfield Thickness on OCT Baseline to 3 Years
Description: as for outcome 6
Time Frame: baseline to 3 years
Population: The study discontinued early. Only subjects with 3 years data are included in 3 year analysis.
Measure: Median (Inter-Quartile Range); unit: Microns
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 111 | 87 | 89
Microns | -158 [-273 to -75] | -103 [-248 to 4] | -114 [-224 to -50]

15. Secondary Outcome: Percentage of Eyes With a Change in Central Subfield Thickness on OCT <250 Microns From Baseline to 3 Years
Description: as for outcome 6
Time Frame: Baseline to 3 years
Population: The study discontinued early. Only subjects with 3 years data are included in 3 year analysis.
Measure: Number; unit: Percentage of Eyes
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Number analyzed (Participants) | 111 | 87 | 89
Percentage of Eyes | 68 | 43 | 51

ADVERSE EVENTS:
Arm/Group | Focal/Grid Laser Photocoagulation | 1mg Intravitreal Triamcinolone | 4 mg Intravitreal Triamcinolone
Serious Adverse Events (participants affected / at risk) | 135/330 | 69/256 | 54/254
Other Adverse Events (participants affected / at risk) | 69/330 | 98/256 | 163/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Focal/Grid Laser Photocoagulation (N=330) | 1mg Intravitreal Triamcinolone (N=256) | 4 mg Intravitreal Triamcinolone (N=254)
Abdominal discomfort (General disorders) | 1 | 0 | 1
Abdominal hernia (General disorders) | 1 | 0 | 0
Abdominal pain (General disorders) | 4 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Allergy to arthropod bite (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 2
Angina unstable (Cardiac disorders) | 2 | 0 | 1
Angioplasty (Vascular disorders) | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 1 | 0
Arteriosclerosis coronary artery (Vascular disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Asbestosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Bladder transitional cell carcinoma (Renal and urinary disorders) | 1 | 0 | 0
Blindness (Eye disorders) | 2 | 0 | 0
Blood count abnormal (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood electrolytes decreased (Blood and lymphatic system disorders) | 1 | 1 | 0
Blood glucose abnormal (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood glucose decreased (Blood and lymphatic system disorders) | 2 | 0 | 1
Blood glucose increased (Blood and lymphatic system disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Breast cancer (Reproductive system and breast disorders) | 2 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Bronchitis viral (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 18 | 4 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Carotid artery occlusion (Vascular disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 4 | 2 | 1
Cerebrovascular accident (Vascular disorders) | 7 | 2 | 1
Chest pain (General disorders) | 9 | 1 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colonoscopy abnormal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colostomy closure (General disorders) | 1 | 0 | 0
Compression fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Convulsion (General disorders) | 1 | 0 | 0
Coronary arterial stent insertion (Vascular disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 0 | 2
Death (General disorders) | 9 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Dehydration (General disorders) | 2 | 0 | 2
Dementia (Psychiatric disorders) | 1 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 2 | 0 | 0
Diabetic coma (Endocrine disorders) | 1 | 1 | 0
Diabetic complications (Endocrine disorders) | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Dialysis (Renal and urinary disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 1 | 0
Dizziness (General disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 2
Endarterectomy (Vascular disorders) | 1 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1
Fall (General disorders) | 1 | 0 | 0
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastric bypass (Gastrointestinal disorders) | 2 | 0 | 0
Gastroenteritis viral (Gastrointestinal disorders) | 2 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal infection (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal injury (Gastrointestinal disorders) | 1 | 1 | 0
Generalised oedema (General disorders) | 2 | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Head injury (General disorders) | 1 | 0 | 0
Headache (General disorders) | 1 | 0 | 1
Heart rate increased (Cardiac disorders) | 1 | 0 | 0
Heart rate irregular (Cardiac disorders) | 2 | 0 | 0
Hernia (General disorders) | 1 | 0 | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Hyperglycaemia (General disorders) | 2 | 1 | 0
Hyperkalaemia (General disorders) | 2 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Hypoglycaemia (General disorders) | 1 | 0 | 0
Hypoxia (General disorders) | 1 | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Intermittent claudication (General disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Kidney infection (Renal and urinary disorders) | 1 | 1 | 0
Knee arthroplasty (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Limb injury (General disorders) | 2 | 1 | 1
Limb operation (Surgical and medical procedures) | 1 | 1 | 0
Localised infection (Infections and infestations) | 5 | 3 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Meniscus lesion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 1 | 0
Metatarsal excision (Surgical and medical procedures) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 16 | 2 | 3
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
oedema (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 2 | 2 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Ovarian cancer (Reproductive system and breast disorders) | 2 | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Pain in extremity (General disorders) | 1 | 1 | 0
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 1
Pneumonia bacterial (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Prostate examination abnormal (Reproductive system and breast disorders) | 1 | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Pulmonary embolism (Vascular disorders) | 1 | 1 | 0
Pulmonary oedema (Vascular disorders) | 1 | 1 | 0
Pulse absent (Cardiac disorders) | 1 | 0 | 0
Rectal haemorrhage (Vascular disorders) | 2 | 0 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 6 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 2 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Renal transplant (Renal and urinary disorders) | 2 | 0 | 1
Renal vessel disorder (Renal and urinary disorders) | 1 | 1 | 0
Rib fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1
Shunt malfunction (General disorders) | 1 | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0
Skin lesion excision (Surgical and medical procedures) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Stent placement (Surgical and medical procedures) | 2 | 0 | 1
Surgical vascular shunt (Surgical and medical procedures) | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tobacco abuse (General disorders) | 1 | 0 | 1
Toe amputation (Surgical and medical procedures) | 5 | 0 | 0
Transient ischaemic attack (Cardiac disorders) | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 2 | 0 | 0
Vascular dementia (Psychiatric disorders) | 1 | 0 | 0
Vertigo (General disorders) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Volvulus (Infections and infestations) | 1 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Focal/Grid Laser Photocoagulation (N=330) | 1mg Intravitreal Triamcinolone (N=256) | 4 mg Intravitreal Triamcinolone (N=254)
Anterior Chamber Cell (Eye disorders) | 1 | 14 | 9
Cataract (Eye disorders) | 38 | 29 | 57
Cataract Cortical (Eye disorders) | 19 | 22 | 32
Cataract Nuclear (Eye disorders) | 13 | 30 | 38
Cataract Operation (Eye disorders) | 14 | 16 | 31
Cataract Subcapsular (Eye disorders) | 29 | 54 | 75
Conjunctival Hemorrhage (Eye disorders) | 7 | 96 | 105
Diabetic Retinopathy (Eye disorders) | 12 | 13 | 5
Dry Eye (Eye disorders) | 10 | 13 | 10
Eye Irritation (Eye disorders) | 2 | 12 | 15
Eye Pain (Eye disorders) | 11 | 28 | 33
Eye Pruritus (Eye disorders) | 9 | 14 | 11
Foreign body in the eye (Eye disorders) | 4 | 61 | 51
Intraocular Pressure increased (Eye disorders) | 14 | 50 | 97
Lacrimation increased (Eye disorders) | 9 | 19 | 16
Maculopathy (Eye disorders) | 23 | 31 | 31
Vision Blurred (Eye disorders) | 36 | 44 | 48
Visual acuity reduced (Eye disorders) | 47 | 40 | 51
Visual disturbance (Eye disorders) | 15 | 23 | 22
Vitreous Detachment (Eye disorders) | 16 | 13 | 7
Vitreous floaters (Eye disorders) | 36 | 92 | 98
Vitrous Hemorrhage (Eye disorders) | 49 | 43 | 32
Anaemia (Blood and lymphatic system disorders) | 21 | 24 | 13
Cardiac Failure Congestive (Cardiac disorders) | 19 | 17 | 14
Dysonoea (General disorders) | 15 | 13 | 16
Headache (General disorders) | 15 | 11 | 20
Hypercholesterolaemia (Blood and lymphatic system disorders) | 11 | 6 | 13
Hypertension (Cardiac disorders) | 17 | 15 | 21
Oedema peripheral (General disorders) | 14 | 13 | 8
Renal failure (Renal and urinary disorders) | 14 | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No